CLINICAL TRIAL: NCT06813885
Title: Evaluation of the Safety and Performance of the TriOSS®: A Prospective Observational Study in Dental Area
Acronym: TriOSSD01
Status: Active, not recruiting | Type: Observational
Sponsor: Bioceramed (Industry)
Collaborators: Egas Moniz - Cooperativa de Ensino Superior, CRL (Other)
Responsible Party: Sponsor
Other Study IDs: TriOSSD01
Record Dates: First submitted 2025-01-29; First posted 2025-02-07 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Bone Augmentation
Keywords: prospective observational clinical study; bone substitute; TriOSS ®; real-world clinical data; efficacy and safety; medical device; reconstructive dental surgeries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to collect real-world clinical data to gather information on the performance and safety of the TriOSS® when used according to its intended purpose and current clinical applications. The results of the clinical study will serve as clinical evidence for the device's clinical evaluation, targeting submission to the new Medical Device Regulation (EU) 2017/745.

DETAILED DESCRIPTION:
TriOSS® is an implantable synthetic calcium phosphate ceramic bone substitute, composed of beta-tricalcium phosphate. The structures composed of this calcium phosphate ceramic material are rapidly osseointegrated due to its chemical composition, which is similar to the mineral phase of the human bone, and due to the interconnected porosity allowing a total vascularization of the implant. Since beta-tricalcium phosphate is more soluble than hydroxyapatite, this material composition enhances and accelerates the bone regeneration process in case of fracture or bone loss. TriOSS® is constituted by the following components: β-tricalcium phosphate, apyrogenic water, dispersing agent, polyurethane foam, and polyvinyl pyrrolidone but most of them don't have a direct contact with the patient.

TriOSS® is gamma sterilized, implantable medical device intended to be use in filling bony voids or gaps of the skeletal system (such as the sinus and alveolar ridge) that are not intrinsic to the stability of the bony structure. These defects may be surgically created defects or osseous defects created from traumatic injury to the bone in adults.

TriOSS® holds CE marking since 2016 and according to rule 8 of Annex VIII of the European Regulation n°2017/745, this product is a class III medical device.

This observational post-market study will collect data relating to standard practice procedures, therefore there are no additional risks or direct benefits associated with participating in this registry for the patient.

This study based on observations of clinical practice aims to collect clinical data to keep up to date the information on the performance and safety of the medical device when used in accordance with its intended use and current clinical applications. The results of the clinical study shall be used as clinical evidence for clinical evaluation of the device aiming submission to the new Medical Device Regulation (EU) 2017/745.

The post-market study is meant to identify and analyse emerging risks, ensure the continued acceptability of the benefit/risk ratio and also identify possible systematic misuse or unauthorized use of the medical device. This protocol does not include any planned new uses, new populations, new materials or design changes.

The results from the prospective observational post-market study will provide an evidence base for assessing the device's performance and safety after its market launch. Detecting real discrepancies in clinical performance between of the medical device early on can offer valuable opportunities to improve device design. This complements the data collected during the pre-market phases, thus improving patient selection. Active surveillance of the safety of medical devices, achieved through the continuous monitoring of vast sources of clinical data, is a priority in the field of medical devices, a requirement of MDR regulation No. 2017/745. This approach is crucial to achieving the objectives set, guaranteeing the safety and efficacy of the devices in circulation.

Patients will be followed as per local standard medical practices of the centre for 2 years.

Clinical data will be collected at 4 points in time: Visit 1 (moment after surgery - baseline and enrolment), Visit 2 (6 months ±3 weeks), Visit 3 (12 months ±30 days) and Visit 4 (23 months ±30 days).

ELIGIBILITY:
Inclusion Criteria:

* Adult males or females (age > 18 years old);
* Patients undergoing reconstructive dental surgeries who meet predefined criteria in Instructions For Use (IFU) of TriOSS®;
* Patients who are able to sign an informed consent form (for data collection);
* Patients who are candidates for bone augmentation procedures in the sinus or alveolar ridge.

Exclusion Criteria:

* Patients who are unable to understand consent and the objectives of the study;
* Signs of local or systemic acute/ active or chronic infections;
* Metabolic affections;
* Severe degenerative diseases, conditions in which general bone grafting is not advisable;
* Implementation sites that allow product migration;
* Conditions which require structural support in the skeletal system;
* Conditions where the implantation site is unstable and not rigidly fixated;
* Sensibility to the implantable materials;
* Known hypersensitivity to the implant material.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients undergoing reconstructive dental surgeries.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Primary Performance Endpoint | moment after surgery; 6 months; 12 months; 23 months.
  Bone consolidation on the surgery site (discrete variable: Yes or No), assessed by X-ray images.
Safety Endpoint | moment after surgery; 6 months; 12 months; 23 months.
  The assessment of Adverse Events (AEs) and device deficiencies (DDs) at least possibly related to TriOSS® during the follow-up period of patients.

SECONDARY OUTCOMES:
Surgeon's Satisfaction survey on the medical device and Technical Success | Visit 1 (moment after surgery - baseline and enrolment)
  Information on the surgeon's satisfaction with the device under study should be collected post-operatively through a general questionnaire. This questionnaire will capture the overall experience of the dentists with the medical device TriOSS®.
2. Quality of life measured through the Oral Health Impact Profile (OHIP-14) Questionnaire | moment after surgery; 6 months; 12 months; 23 months.
  QoL will be assessed during the patients' follow-up period. The final results will be categorized as often affected (if they answer 3 or 4 on at least one of the OHIP-14 questions) or little affected (0, 1 or 2 on all items).

CONTACTS AND LOCATIONS:
Locations (1):
- Egas Moniz School of Health and Science, Caparica, Lisbon District, Portugal

IPD SHARING:
Plan to Share IPD: No